CLINICAL TRIAL: NCT00117663
Title: A Population-Based Randomized Trial to Assess the Effects of Short-Term Cessation of Hormone Replacement Therapy (HRT) on Mammography Assessments and Breast Density
Brief Title: Radiologic Evaluation and Breast Density (READ)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DAMD17-03-1-0447
Record Dates: First submitted 2005-06-30; First posted 2005-07-08 (Estimated); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: Randomized controlled trial; Mammography; health care setting; hormone replacement therapy; breast density; mammography performance; Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No Hormone Suspension (No Intervention): No hormone suspension prior to screening mammogram
- 1 month hormone suspension (Active Comparator): discontinuation of hormone therapy for 1 month prior to screening mammogram.
  Interventions: Other: temporary discontinuation of hormone therapy for 1 month
- 2 month hormone suspension (Active Comparator): discontinuation of hormone therapy for 2 months prior to screening mammogram.
  Interventions: Other: temporary discontinuation of hormone therapy for 2 months

INTERVENTIONS:
Other: temporary discontinuation of hormone therapy for 1 month — temporary discontinuation of hormone replacement therapy for 1 month prior to screening mammogram.
  Arms: 1 month hormone suspension
Other: temporary discontinuation of hormone therapy for 2 months — temporary discontinuation of hormone replacement therapy for 2 months prior to screening mammogram
  Arms: 2 month hormone suspension

SUMMARY:
The purpose of this study is to determine whether cessation of hormone replacement therapy for one or two months before a screening mammogram will improve its performance by decreasing breast density.

DETAILED DESCRIPTION:
This randomized, controlled trial is designed to test whether short-term (1-2 months) HRT cessation will sufficiently lower breast density to decrease the proportion of women who receive a recommendation for additional evaluation following a screening mammogram, and to examine whether there is a trend by duration of cessation. The study is being conducted at Group Health Cooperative, a managed health care organization in western Washington State with an organized breast cancer screening program. We are recruiting 1,500 women and will randomize women to one of three HRT arms: 1) cessation two months before the screening mammogram; 2) cessation one month before; and 3) continued HRT use. We are using a computer-assisted method to measure mammographic breast density continuously. Mammography recall rates are being determined from an expert radiologist review of the mammograms, blinded to HRT status.

ELIGIBILITY:
Inclusion Criteria:

* 1 or more prior screening mammograms at Group Health Cooperative within the past 2 years
* Currently taking HRT
* Taking HRT at prior screening mammogram
* Due for a screening mammogram

Exclusion Criteria:

* BI-RADS breast density of 1 (entirely fat)
* Previous cardiovascular events (heart surgery, catheterization, stent bypass, angioplasty, stroke, DVT)
* Previous breast cancer
* History of breast implants
* Breast reduction since last mammogram
* Mastectomy
* History of using Tamoxifen or Raloxifene
* Declined contact or use of data for research

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1704 (Actual)
Dates: Start 2004-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana SM Buist, Ph.D., Principal Investigator — Kaiser Permanente
Locations (1):
- Group Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lowry SJ, Aiello Bowles EJ, Anderson ML, Buist DS. Predictors of breast density change after hormone therapy cessation: results from a randomized trial. Cancer Epidemiol Biomarkers Prev. 2011 Oct;20(10):2309-12. doi: 10.1158/1055-9965.EPI-11-0629. Epub 2011 Aug 3. PMID 21813728
- [Derived] Newton KM, Anderson ML, Reed SD, Bowles EJ, Buist DS. Factors associated with non-compliance with hormone therapy cessation before screening mammography. Climacteric. 2011 Apr;14(2):268-74. doi: 10.3109/13697137.2010.520172. Epub 2010 Oct 27. PMID 20979462
- [Derived] Aiello Bowles EJ, Anderson ML, Reed SD, Newton KM, Fitzgibbons ED, Seger D, Buist DS. Mammographic breast density and tolerance for short-term postmenopausal hormone therapy suspension. J Womens Health (Larchmt). 2010 Aug;19(8):1467-74. doi: 10.1089/jwh.2009.1681. PMID 20575711
- [Derived] Reed SD, Buist DS, Anderson ML, Bowles EJ, Fitzgibbons D, Seger D, Newton KM. Short-term (1-2 mo) hormone therapy cessation before mammography. Menopause. 2009 Nov-Dec;16(6):1125-31. doi: 10.1097/gme.0b013e3181a5ce60. PMID 19455069
- See also: Link for patients — http://www.ncbi.nlm.nih.gov/pubmed/19487707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1704 women age 45 to 80 years who used hormone therapy at their most recent screening (index) mammography, were due for screening (study) mammography, and were still using hormone therapy.
Groups:
- 1 Month Hormone Suspension: 1 month of hormone suspension prior to screening mammogram
Period: Overall Study
Arm/Group | No Hormone Suspension | 1 Month Hormone Suspension | 2 Month Hormone Suspension
Started | 567 | 570 | 567
Completed | 542 | 478 | 451
Not Completed | 25 | 92 | 116

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Hormone Suspension | 1 Month Hormone Suspension | 2 Month Hormone Suspension | Total
Number analyzed (Participants) | 567 | 570 | 567 | 1704
Age, Customized [Number; unit: participants]
  45 - 80 years | 567 | 570 | 567 | 1704
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 567 | 570 | 567 | 1704
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 567 | 570 | 567 | 1704

OUTCOME MEASURES:

1. Primary Outcome: Mammogram Recall for Additional Imaging
Description: Mammography recall was defined as any assessment requiring additional imaging or evaluation of either breast (BI-RADS assessment of 0 for either or both breasts)(30) determined exclusively from the study radiologists' interpretation.
Time Frame: 4 years
Measure: Number (95% Confidence Interval); unit: percentage of women recalled
Groups:
- No Hormone Suspension: Hormone Replacement Therapy (HRT) was not interrupted prior to mammogram in this arm.
- 1 Month Hormone Suspension: Hormone Replacement Therapy (HRT) was suspended for 1 month prior to mammogram then resumed.
- 2 Month Hormone Suspension: Hormone Replacement Therapy (HRT) was interrupted for 2 months prior to mammogram then resumed in this arm.
Arm/Group | No Hormone Suspension | 1 Month Hormone Suspension | 2 Month Hormone Suspension
Number analyzed (Participants) | 542 | 478 | 451
percentage of women recalled | 11.3 [8.7 to 14.2] | 12.3 [9.5 to 15.6] | 9.8 [7.2 to 12.9]

2. Primary Outcome: Mammographic Breast Density
Description: Breast density (Mean, SE) and Change in Breast density by Randomization Group
Time Frame: 4 years
Measure: Mean (Standard Error); unit: Change in % dense
Arm/Group | No Hormone Suspension | 1 Month Hormone Suspension | 2 Month Hormone Suspension
Number analyzed (Participants) | 541 | 478 | 452
Change in % dense | 0.1 (0.3) | -0.9 (0.3) | -1.5 (0.4)

ADVERSE EVENTS:
Groups:
- 2 Month Hormone Suspension: 2 months of hormone suspension prior to screening mammogram
Arm/Group | No Hormone Suspension | 1 Month Hormone Suspension | 2 Month Hormone Suspension
Serious Adverse Events (participants affected / at risk) | 5/527 | 1/462 | 2/443
Other Adverse Events (participants affected / at risk) | 13/527 | 6/462 | 0/443
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Hormone Suspension (N=527) | 1 Month Hormone Suspension (N=462) | 2 Month Hormone Suspension (N=443)
Myocardial Infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Stroke (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Hormone Suspension (N=527) | 1 Month Hormone Suspension (N=462) | 2 Month Hormone Suspension (N=443)
Breast Cancer (Reproductive system and breast disorders) | 3 (3) | 0 (0) | 0 (0)
Atypical Chest Pain (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Other adverse event (General disorders) | 8 (8) | 6 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes